CLINICAL TRIAL: NCT02185066
Title: Phase 1 Study to Compare the Safety, Pharmacokinetic Profiles of CJ-30056 and Lipitor/Glucophage XR
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_ATM_103
Record Dates: First submitted 2014-07-07; First posted 2014-07-09 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Single-dose crossover
  1. Reference: Atorvastatin 20mg and Metformin XR 500mg
  2. Test: CJ-30056 20/500mg
  Once daily Oral administration with 7days of washout period
  Interventions: Drug: Atorvastatin 20mg and Metformin XR 500mg (Reference); Drug: CJ-30056 20/500mg (Test)
- Group 2 (Experimental): Single-dose crossover
  1. Test: CJ-30056 20/500mg
  2. Reference: Atorvastatin 20mg and Metformin XR 500mg
  Once daily Oral administration with 7days of washout period
  Interventions: Drug: Atorvastatin 20mg and Metformin XR 500mg (Reference); Drug: CJ-30056 20/500mg (Test)

INTERVENTIONS:
Drug: Atorvastatin 20mg and Metformin XR 500mg (Reference) — Group 1 receives Atorvastatin 20mg and Metformin XR 500mg first, then CJ-30056 second, with at 7-day wash-out period in between.
  Group 2 receives CJ-30056 first, then Atorvastatin 20mg and Metformin XR 500mg second, with 7-day wash-out period in between.
Drug: CJ-30056 20/500mg (Test) — Group 1 receives Atorvastatin 20mg and Metformin XR 500mg first, then CJ-30056 second, with at 7-day wash-out period in between.
  Group 2 receives CJ-30056 first, then Atorvastatin 20mg and Metformin XR 500mg second, with 7-day wash-out period in between.

SUMMARY:
This study is designed to evaluate safety and pharmacokinetic properties of the two treatments, the administration of CJ-30056 and the co-administration of atorvastatin and metformin XR, in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Willing to adhere to protocol requirements and sign a informed consent form
2. Male volunteers in the age between 19 and 55 years old and have the weight range is not exceed ±20% of ideal weight
3. Subjects with no history of any significant chronic disease
4. Judged to be in good health on the basis of their vital sign, ECG, physical exam and routine laboratory data

Exclusion Criteria:

1. Use of barbital inducer or inhibitor medication within the 4 weeks before dosing
2. Symptom of an acute illness within 4 weeks prior to drug administration
3. History of clinically significant hepatic, renal, gastrointestinal diseases which might significantly interfere with ADME
4. History of surgery except or gastrointestinal diseases which might significantly change absorption of medicines
5. History of clinically significant allergies including drug allergies
6. History of clinically significant allergies about atorvastatin or metformin
7. Subjects who have ever or have plan to do intravenous injection of contrast medium (intravenous urography, intravenous cholangiography, computed tomography using contrast medium) within 28 days prior to drug administration
8. History of myopathy
9. Clinical laboratory test values are outside the accepted normal range

   * AST or ALT >1.25 times to normal range
   * Total bilirubin >1.5 times to normal range
   * e-GFR <90 mL/min
10. History of drug, caffein(caffein > 5 cups/day), smoking (cigarette > 10/day) or alcohol abuse(alcohol > 30 g/day)or Subjects who have ever drink within 7 days prior to drug administration
11. Special diet known to interfere with the absorption, distribution, metabolism or excretion of drugs (especially, consumption of grapefruit juice) within 7 days prior to drug administration
12. Donated blood within 60 days prior to dosing
13. Participated in a previous clinical trial within 60 days prior to dosing
14. Use of any other medication, including herbal products, within 10 days before dosing
15. Subjects considered as unsuitable based on medical judgement by investigators

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of Atorvastatin | Upto 36 hours
Maximum plasma concentration (Cmax) of Metformin | Upto 24 hours
Area Under the plasma concentration-time Curve (AUC0-t) of Atorvastatin | Upto 36 hours
Area Under the plasma concentration-time Curve (AUC0-t) of Metformin | Upto 24 hours

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of 2-OH-atorvastatin | Upto 36 hours
Area Under the plasma concentration-time Curve (AUC0-t) of 2-OH-atorvastatin | Upto 36 hours
CL/F of Atorvastatin and Metformin | Upto 36 hours
Vd/F of Atorvastatin and Metformin | Upto 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: Jong-lyul Ghim, MD. PhD, Principal Investigator — Inje University
Locations (1):
- Inje University Busan Paik Hospital, Busan, South Korea